CLINICAL TRIAL: NCT00016601
Title: An Open-Label, Non-Randomized Study of Pharmacokinetic Interactions Between Depo-Medroxyprogesterone Acetate (DMPA, Depo-Provera) and Selected Protease Inhibitor (PI) and Nonnucleoside Reverse Transcriptase Inhibitor (NNRTI) Therapies Among HIV-Infected Women
Brief Title: Depo-Medroxyprogesterone Acetate (DMPA, Depo-Provera) Use With Certain Anti-HIV Drugs in HIV-Infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Purpose: Treatment
Other Study IDs: A5093; ACTG A5093
Record Dates: First submitted 2001-05-18; First posted 2001-08-31 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Delayed-Action Preparations; Drug Interactions; Drug Therapy, Combination; Nevirapine; HIV Protease Inhibitors; Ritonavir; Indinavir; Nelfinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Pharmacokinetics; Medroxyprogesterone 17-Acetate; efavirenz
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; Nelfinavir; efavirenz; Nevirapine; Medroxyprogesterone Acetate

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Efavirenz
Drug: Nevirapine
Drug: Medroxyprogesterone acetate

SUMMARY:
The purpose of this study is to look at the level of depo-medroxyprogesterone acetate (DMPA or Depo-Provera) in the blood to see if is affected by certain anti-HIV drugs (nelfinavir [NFV], efavirenz [EFV], indinavir [IDV] in combination with ritonavir [RTV], and nevirapine [NVP]). This study will also look at the levels of these anti-HIV drugs to see if they are affected by DMPA.

DMPA is a hormonal birth control method that is given as an injection. It is not known if taking DMPA together with anti-HIV drugs changes the amount of DMPA and/or the amount of anti-HIV drugs in the blood. If higher levels of DMPA occur, side effects may increase. If lower levels of anti-HIV drugs occur, the drugs may become less effective against HIV. This study will look at the levels of anti-HIV drugs and DMPA in the blood when these medications are used together.

DETAILED DESCRIPTION:
DMPA, an injectable depot formulation of medroxyprogesterone (MPA), is a commonly used form of "progestin-only" contraception. Information is limited on the specific P450 isozymes that metabolize MPA; however, it appears that CYP3A4 is 1 pathway of hepatic clearance. Drugs known to be inhibitors of the CYP3A4 pathway (such as protease inhibitors [PIs]) may lead to elevated concentrations of MPA. Secondly, MPA given as DMPA injections has been shown to induce the activity of CYP3A4 by 25 percent. It is possible that this action may result in enhanced clearance of the substrates of CYP3A4, including PIs and nonnucleoside reverse transcriptase inhibitors (NNRTIs), which in turn may result in reduced drug exposure and possible ARV failure. This study is designed to address the lack of information on potential interactions between PIs or NNRTIs and DMPA.

Patients are enrolled into 1 of 5 arms based on their current ARV regimen:

Arm A (control group): No current ARVs or receiving nucleoside reverse transcriptase inhibitors (NRTIs) only.

Arm B: NFV (1250 mg bid or 750 mg tid) in combination with NRTIs. Arm C: EFV (600 mg qd) in combination with NRTIs. Arm D: IDV (800 mg bid) and RTV (100 mg bid or 200 mg bid) in combination with NRTIs.

Arm E: NVP (200 mg bid) in combination with NRTIs. Acceptable NRTIs and any fixed combination of these medications include: zidovudine (ZDV), lamivudine, didanosine, stavudine (d4T), zalcitabine, and abacavir; concurrent therapy using ZDV and d4T is not allowed. ARV therapy is not provided by this study. One dose of DMPA is provided to all patients at entry (Day 0) and an optional dose of DMPA will be available at the final visit (Week 12) for those who are interested in continuing with DMPA outside of the protocol and who do not experience adverse events from the first DMPA injection. Patients in Arms B, C, D, and E have intensive pharmacokinetic sampling done at entry and at Week 4 to measure ARV levels. All patients have blood tests at Weeks 2, 4, 6, 8, 10, and 12 to measure levels of DMPA and progesterone. In addition, tests to monitor HIV-1 RNA levels, CD4 and CD8 counts, hematology, blood chemistries, and liver function are performed periodically.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Have plasma HIV-1 RNA (level of HIV in the blood) below 10,000 copies/ml within 30 days before study entry.
* Had their last menstrual period (LMP) less than 35 days before study entry.
* Have serum follicle-stimulating hormone below 40 MIU/ml if their LMP occurred more than 35 days before study entry.
* Have been on the same anti-HIV drugs for at least 30 days before study entry, if taking anti-HIV drugs. If not taking anti-HIV drugs, patients must have been told about anti-HIV drugs within the 3 months before study entry and have chosen not to take them now or in the future.
* Intend to continue on their anti-HIV drugs, if taking them, for at least 3 months after study entry.
* Have a CD4 cell count above 200 cells/mm3 if taking anti-HIV drugs, or a CD4 cell count above 350 cells/mm3 if not taking anti-HIV drugs, within 30 days before study entry.
* Have not had menopause (change of life) and have a normal reproductive system.
* Have not had any infections or AIDS-related diseases requiring drugs within 14 days before study entry.
* Are 13 years of age or older.
* Are female.
* Have a negative pregnancy test within 30 days before study entry.
* Agree to avoid becoming pregnant for the entire study. If sexually active, agree to use at least 1 barrier method of birth control (male or female condom with or without spermicide [a cream or gel that kills sperm] or diaphragm or cervical cap with spermicide) while receiving DMPA in this study.
* Have consent of a parent or guardian if under 18 years of age.
* Weigh at least 40 kg (88 lbs) and are within a certain range of their ideal body weight.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have taken anti-HIV drugs within 30 days before study entry but have chosen not to take them.
* Are taking only 1 NRTI.
* Are taking anti-HIV drugs other than those listed in the treatment groups, including tenofovir, amprenavir, and lopinavir/ritonavir, or have taken tenofovir, amprenavir, or lopinavir/ritonavir within 30 days before study entry.
* Have taken ZDV and d4T together within 30 days before study entry.
* Are not able to take the anti-HIV drugs properly while on the study, in the opinion of the investigator.
* Are allergic to DMPA, MPA, or any of the other ingredients in DMPA.
* Have received DMPA within 180 days before study entry.
* Have received other hormones (Provera, oral contraceptives, hormonal replacement therapy, or anabolic drugs [e.g., nandrolone decanoate, megestrol acetate]) within 30 days before study entry.
* Are taking any of the following: amiodarone, astemizole, bepridil, buspirone, carbamazepine, cimetidine, cisapride, clarithromycin, cyclosporine, dihydroergotamine, diltiazem, ergotamine, erythromycin, flecainide, glucocorticoids, grapefruit juice, St. John's wort, itraconazole, ketoconazole, lovastatin, midazolam, nefazodone, phenobarbital, phenytoin, pimozide, pioglitazone, propafenone, propofol, quinidine, rifabutin, rifampin, rosiglitazone, simvastatin, tacrolimus, terfenadine, ticlopidine, triazolam, or verapamil.
* Have taken any of the following drugs within 30 days before study entry: amiodarone, astemizole, bepridil, buspirone, carbamazepine, cisapride, clarithromycin, cyclosporine, dihydroergotamine, ergotamine, erythromycin, flecainide, glucocorticoids, St. John's wort, itraconazole, ketoconazole, lovastatin, midazolam, nefazodone, phenobarbital, phenytoin, pimozide, pioglitazone, propafenone, propofol, quinidine, rifabutin, rifampin, rosiglitazone, simvastatin, tacrolimus, terfenadine, ticlopidine, or triazolam.
* Have started, stopped, or changed doses, within 30 days before study entry, of certain drugs including: benzodiazepines, except midazolam and triazolam; bupropion; calcium channel blockers, except diltiazem and verapamil; fluconazole; lipid-lowering drugs except pravastatin (i.e., atorvastatin, cerivastatin, and fluvastatin, but not lovastatin and simvastatin); isoniazid; mexiletine; zaleplon; and zolpidem. The patient can, however, remain on stable doses of these drugs during the study.
* Are receiving methadone maintenance treatment for less than 60 days before study entry.
* Are breast-feeding.
* Have had a baby within 30 days before study entry.
* Have had their uterus or both ovaries removed.
* Abuse drugs or alcohol.
* Cannot stop drinking alcohol 1 day before and during the testing at entry and at Week 4.
* Have had a change in smoking habits within 6 weeks before study entry. Patients may have either stopped or started smoking more than 6 weeks before study entry.
* Have cancer of the reproductive system, vaginal bleeding of unknown cause, thyroid problems, liver tumors, or serious eye problems at any time before study entry.
* Are taking investigational drugs without approval of the protocol chair.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76
Dates: Start 2001-06; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Cohn, Study Chair
Locations (32):
- United States (31):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Mt Sinai Hosp Med Ctr / Dept of Pediatrics, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Childrens Memorial Hosp (Pediatric), Chicago, Illinois
  - The Univ of Chicago Childrens Hosp, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Methodist Hosp of Indiana / Life Care Clinic, Indianapolis, Indiana
  - Wishard Hosp, Indianapolis, Indiana
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland, Institute of Human Virology, Baltimore, Maryland
  - Boston Med Ctr (Pediatric), Boston, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Beth Israel Med Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Community Health Network, Inc, Rochester, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve Univ, Cleveland, Ohio
  - MetroHealth Med Ctr, Cleveland, Ohio
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Texas Galveston, Galveston, Texas
  - Univ of Washington, Seattle, Washington
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- San Juan City Hosp, San Juan, Puerto Rico

REFERENCES:
- [Result] Watts DH, Park JG, Cohn SE, Yu S, Hitti J, Stek A, Clax PA, Muderspach L, Lertora JJ. Safety and tolerability of depot medroxyprogesterone acetate among HIV-infected women on antiretroviral therapy: ACTG A5093. Contraception. 2008 Feb;77(2):84-90. doi: 10.1016/j.contraception.2007.10.002. Epub 2007 Dec 21. PMID 18226670